CLINICAL TRIAL: NCT03797170
Title: Design of New Personalized Therapeutic Approaches for Diffuse Large B-cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Pier Luigi Zinzani, Full Professor, MD (Hematologist), University of Bologna
Other Study IDs: Oncopassport; RF-2016-02363730 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2018-12-19; First posted 2019-01-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: RCHOP; first line; microbiota; response; disease control; therapy toxicity
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Gut microbiota
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gut microbiota samples — Gut microbiota analysis from diagnosis to follow up after first line-chemo-immuntherapy

SUMMARY:
In Europe diffuse large B-cell lymphoma (DLBCL) is a rare disease whereas in Italy it is not. Approximately 40% of DLBCL patients has refractory disease or will relapse after initial response. In onco-hematology, a role for gut microbiota (GM) in mediating immune activation in response to chemotherapy, has been suggested. In this scenario, the Investigators hypothesized that GM could play an important role in DLBCL prognosis and response to treatment, establishing a connection between lifestyle and clinical response. The project is aimed to the study of the functional GM layout in association with specific patterns of treatment response in de novo DLBCL undergoing standard first line chemo-immunotherapy. Results may build the scientific basis to design new and personalized intervention strategies (both in treatment approach and in life-style recommendations), to enhance clinical response and reduction of disease refractoriness through modulation of the gut microbial ecosystem.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients affected by histologically confirmed diffuse large B-cell lymphoma
3. Patients amenable for therapy with RCHOP (RCHOP is the standard first line therapy for DLBCL and it scheduled regardless of participation in present study).
4. Patients must provide written informed consent.

Exclusion Criteria:

1. Concomitant second malignancy, other than lymphoma.
2. Previous anti-lymphoma therapy.
3. Pregnancy or breastfeeding.
4. Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by diffuse large B-cell lymphoma (DLBCL) undergoing therapy with front-line R-CHOP (rituximab-cyclophosphamide, doxorubicin, vincristine, prednisone).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2023-07-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
GM dysbiosis assessment (bacterial DNA of gut microbiota in all patients) | 18 months
  * dysbiosis index: the dysbiosis index relies on the calculation of the weighted ratio between health-promoting and disease-associated GM components
  * relative abundance of GM biomarkers of an eubiotic GM state: all GM dysbiotic states share a common feature, i.e. the depletion of strategic health-promoting GM components such as Faecalibacterium prausnitzii and Lachnospiraceae. Thus, a GM dysbiotic state is determined by the assessment of a reduction of the abundance of these GM biomarkers below the thresholds characteristic of an eubiotc GM state.

SECONDARY OUTCOMES:
Response to therapy | 2 years
  Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. when the PET scan was positive before therapy, a post-treatment residual mass of any size is permitted as long as it is PET negative and all lymph nodes and nodal masses must have regressed on CT to normal size ( 1.5 cm in their greatest transverse diameter for nodes 1.5 cm before therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi L Zinzani, Professor, Principal Investigator — Institute of Hematology "L. e A. Seràgnoli", University of Bologna
Locations (2):
- Italy (2):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola, FC
  - Institute Of Hematology "Seràgnoli", Bologna

IPD SHARING:
Plan to Share IPD: Undecided